CLINICAL TRIAL: NCT02301598
Title: Femtosecond Laser-assisted Anterior Lamellar Keratoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The S.N. Fyodorov Eye Microsurgery State Institution (Other Government)
Responsible Party: Principal Investigator, Alexey Pashtaev, Alexey Pashtaev MD, PhD, The S.N. Fyodorov Eye Microsurgery State Institution
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FS-1
Record Dates: First submitted 2014-11-20; First posted 2014-11-26 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Keratoconus; Corneal Opacity
Keywords: femtosecond laser; anterior lamellar keratoplasty; atomic-force microscopy
MeSH Terms: conditions — Keratoconus; Corneal Opacity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FS-ALK (Experimental): Femtosecond laser-assisted maximum thickness anterior lamellar keratoplasty (FS-ALK) was performed for 11 eyes of 11 patients with advanced keratoconus and 2 eyes of 2 patients with superficial corneal scattering.
  Interventions: Procedure: FS-ALK (Femtolaser-assisted anterior lamellar keratoplasty)

INTERVENTIONS:
Procedure: FS-ALK (Femtolaser-assisted anterior lamellar keratoplasty) — The procedure was a non-penetrating transplantation of 80% thickness corneal graft
  Other Names: Femto-ALK

SUMMARY:
The purpose of the study is evaluating safety and clinical efficiency of full femtosecond laser-assisted anterior lamellar keratoplasty (FS-ALK) for curing patients with keratoconus and corneal opacities

DETAILED DESCRIPTION:
Keratoplasty is the most widely spread tissue transplantation procedure. Although penetrating keratoplasty (PKP) is still commonly used for curing corneal dystrophy and opacities of different genesis, lamellar techniques provide significant advantages in terms of safety and predictability.

Al in all 13 FS-ALK procedures were performed for 11 eyes with advanced keratoconus and 2 eyes with superficial corneal scattering Before and after surgery uncorrected visual acuity (UCVA), best spectacle-corrected visual acuity (BSCVA), postoperative astigmatism, endothelial cell loss, central cornea thickness, residual recipient's tissue thickness, corneal hysteresis (CH) and corneal resistance factor (CFR) were evaluated . At 1-year follow-up Confoscan investigation of donor-recipient interface was performed.

All FS-ALK procedures were performed with Intralase FS 60kHz femtosecond laser in a following way. At first a 80% thickness corneal graft was prepared. Then maximum thickness recipients corneal dissection was performed according to OCT (optical coherence tomography) data and superficial tissue was removed. Transplant was fixed in a resulted bed by continuous suture.

ELIGIBILITY:
Inclusion Criteria:

* Advanced keratoconus or stromal corneal scattering
* Normal endothelial cell density

Exclusion Criteria:

* Acute keratoconus in the anamnesis
* Low endothelial cell density
* Age under 18 years

Ages: 18 Years to 52 Years | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Mean endothelial cell loss | 12 months after surgery
Mean postoperative astigmatism | 12 months after surgery
UCVA (uncorrected visual acuity) | 12 months after surgery
BSCVA (best spectacle-corrected visual acuity) | 12 months after surgery

SECONDARY OUTCOMES:
Corneal hysteresis | 12 months after surgery
  Evaluation of biomechanical qualities of the cornea
Corneal resistance factor | 12 months after surgery
  Evaluation of biomechanical qualities of the cornea
Central corneal thickness | 12 months after surgery
  measured by OCT (optical coherence tomography - Optovue)
Residual recipient's tissue thickness | 12 months after surgery
  measured by OCT (optical coherence tomography - Optovue)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Malyugin, MD,PhD,prof., Study Director — The S.N. Fedorof Federal State Institution